CLINICAL TRIAL: NCT03382132
Title: momHealth: Multiple Health Behavior Change Intervention in Teen Pregnancy & Parenting Using Mobile Technology
Acronym: momHealth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00141254; R21HD088913-01A1 (NIH)
Record Dates: First submitted 2017-12-13; First posted 2017-12-22 (Actual); Last update posted 2020-09-03 (Actual); Status verified 2020-09

CONDITIONS: Health Behavior
MeSH Terms: conditions — Health Behavior | interventions — Standard of Care

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- momHealth (Experimental): Participants will receive support and information via the momHealth program.
  Interventions: Behavioral: momHealth
- Control (Active Comparator): Participants will receive the normal support they would normally receive if they were not in a study.
  Interventions: Behavioral: Standard of Care

INTERVENTIONS:
Behavioral: momHealth — Mobile health program delivered via an iPad. Program delivers information and support related to breastfeeding education, Ten Steps of the Baby Friendly Hospital Initiative, healthy eating and active living topics, and depression prevention information.
  Arms: momHealth
Behavioral: Standard of Care — Participants will receive standard health care via their prenatal provider, including routine prenatal education and postpartum support.
  Arms: Control

SUMMARY:
The purpose of this study is to find out if information and support provided with a mobile-delivered (via iPad) momHealth Teen Pregnancy Program can promote healthy choices and behaviors during and after pregnancy.

DETAILED DESCRIPTION:
This is a RCT to pilot test an innovative multiple health behavior intervention to influence three areas of health for pregnant and parenting adolescents: breastfeeding, healthy eating/active living, and depression prevention. Intervention and control groups will be compared in the main outcomes of the study (see 4.2.c. and 4.3). Beginning in the last eight weeks of pregnancy and extending to one month after giving birth, we use mobile health technology (e.g., iPad minis) to deliver multi-media educational modules, text-messaging, virtual home visits with professionals using secure televideo, and real-time peer group support over televideo. At birth, five weeks, and three months after giving birth, effectiveness of the program outcomes will be assessed and compared to a usual care control group and include breastfeeding/infant-feeding practices; healthy eating and physical activity; and depressive symptoms. This is the first known study to address these multiple behaviors simultaneously with pregnant and parenting adolescent women.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant females
* English-speaking
* Giving birth to first child
* Intending to keep the newborn
* Access to a telephone
* 27-31 weeks gestation
* Low-risk pregnancy

Exclusion Criteria:

* Multiple gestation pregnancy
* High-risk pregnancy
* Women with active untreated mental health conditions such as affective disorder, substance use disorder, anxiety disorder (excluding simple phobia), or psychosis

Ages: 15 Years to 20 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes
Enrollment: 78 (Actual)
Dates: Start 2017-09-20 (Actual); Primary Completion 2020-05-25 (Actual); Study Completion 2020-08-30 (Actual)

PRIMARY OUTCOMES:
Duration of breastfeeding | Month 3
  Number of days out to 3 months postpartum of any breastfeeding.
Consumption of "red" foods per day | Change from Baseline to Month 3
  Measure will be assessed using the Automated Self-Administered 24-hour Recall™ (ASA24™). Participants will provide information on food eaten through an online site and accessed with an individualized link.
Minutes of moderate to vigorous physical activity per week | Change from Baseline to Month 3
  Measure will be assessed using ActiGraph Physical Activity Monitors.
Change in depressive symptoms | Month 3
  Assessed using the Edinburgh Postnatal Depression Scale (EPDS), a 10-item questionnaire. Each question response is coded from 0 to 3. Scores can range from a minimum of 0 to a maximum of 30. A score of 10 or greater detects a major depressive disorder with sensitivity.
Rate of any and exclusive breastfeeding | Month 3
  Self-report data on breastfeeding continuation, either wholly or partially, out to 3 months postpartum.

CONTACTS AND LOCATIONS:
Overall Officials: Karen Wambach, PhD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States